CLINICAL TRIAL: NCT02836301
Title: Optimizing Educational Video Designs to Improve Minority Organ Donor Registration - Aim 2 Randomized Trial Comparing Testimonials Versus Documentary Videos
Brief Title: RCT- Comparing Testimonial Versus Documentary Organ Donation Video Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16-00454
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Organ Donation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Testimonials-Uplifting (Active Comparator): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Control ending - Uplifting
- Testimonials-Negative (Active Comparator): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Negative Consequences Ending
- Testimonials-Unresolved (Active Comparator): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Unresolved Ending
- Documentary-Uplifting (Experimental): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Control ending - Uplifting
- Documentary-Negative (Experimental): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Negative Consequences Ending
- Documentary-Unresolved (Experimental): 2x3 matrix for the RCT comparing the control genre of only testimonials (G0) versus the experimental genre (G1) of a documentary with live footage along with the testimonials. The story ending (E) will serve as the cofactor.
  Interventions: Behavioral: Unresolved Ending

INTERVENTIONS:
Behavioral: Control ending - Uplifting — The control ending is emotionally uplifting. In this video, the decedent previously registered as an organ donor through online registration and discussed his decision with family. The scene cuts to the family affirming the deceased's wish. In the next scene, the donor family and recipient meet for the first time, ending with a plea from both parties for viewers to register for donation.
  Arms: Documentary-Uplifting; Testimonials-Uplifting
Behavioral: Negative Consequences Ending — A sad ending where the decedent did not register or discuss their position with family; family is asked to consider donation as an option, but they do not agree. The patient with kidney failure misses the window of opportunity, and the final scene is of both families grieving at their respective family members' grave plots…a missed opportunity.
  Arms: Documentary-Negative; Testimonials-Negative
Behavioral: Unresolved Ending — In this ending, the team checks for registration status, and while searching, the scene cuts to physicians discussing the death with family and whether they might consider preservation and organ donation. The video then cuts to the potential recipient and family hoping for a kidney transplant before it is too late. The story ends without resolution, leaving viewers to contemplate how they might respond in the same situation
  Arms: Documentary-Unresolved; Testimonials-Unresolved

SUMMARY:
Investigators will evaluate organ donation educational videos with a 2x3 single blinded Randomized Control Trial (RCT) in partnership with our 26 Latino Owned Barbershops (LOBs). The testimonial video about Uncontrolled Donation after Circulatory Determination of Death (uDCDD) with an uplifting ending will serve as control. Experimental videos may include live uDCDD footage, differing endings, or combinations. Video production will be informed by the entertainment education model and produced with experts including an Academy Award winning filmmaker. The primary outcome is whether participants immediately enroll in the NY State Organ Donor Registry (either online or by our RA mailing in the official form with prepaid postage). Investigators hypothesize that each video will induce differences in registration compared to the control and that there is an interaction effect with video genre and story outcome.

ELIGIBILITY:
Inclusion Criteria:

* Dominican and Puerto Rican Latinos.
* Participants who pefer to speak Spanish.
* Participants who reside locally in NYC, New Jersey, or Connecticut, (tri-state area) for at least four weeks (28 days) in a year.
* Participants able to understand the verbal consent process.

Exclusion Criteria:

* Persons who are visually impaired and are unable to watch the videos.
* Persons who are hearing impaired and are unable to hear the audio on the videos.
* Persons who are cognitively impaired and thus are unable to provide consent to register for organ donation by signing the New York State Organ Donor Registry application.
* Persons who self-report to be registered in the New York State Organ Donor Registry.
* Persons who previously are enrolled in this randomized controlled trial.
* Persons psychologically unfit or who refuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1440 (Actual)
Dates: Start 2015-05-21 (Actual); Primary Completion 2017-07-15 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
RA Assisted and Observed Immediate Registration | 1 Day

SECONDARY OUTCOMES:
Confirmed Registration NYS DOH aggregate data by video group | 1 Day
Number pf participants who viewed "How To Register" Video | 1 Day
  RA assisted / observed
Number of participants who accepted Information/ Registry Forms | 1 Day
Organ Donation Beliefs (ODBI) Questionnaire | 1 Day
Emotional State (PANAS-CAT) Questionnaire | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wall, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wall SP, Castillo P, Shuchat Shaw F, Norman E, Martinez-Lopez N, Lopez-Rios M, Paulino H, Homer B, Plass JL, Ravenell JE. Including Medical Footage and Emotional Content in Organ Donation Educational Videos for Latinx Viewers. Health Educ Behav. 2022 Jun;49(3):424-436. doi: 10.1177/10901981211022240. Epub 2021 Jul 12. PMID 34253089